CLINICAL TRIAL: NCT05341700
Title: The Effect of Impact Loading on Bone Biomarkers in Energy-Restricted Female Runners
Brief Title: Impact Loading Effect on Bone Biomarkers in Female Runners
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Polytechnic Institute and State University (Other)
Responsible Party: Principal Investigator, Dawnine Enette Larson-Meyer, Professor, Virginia Polytechnic Institute and State University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 22-168
Record Dates: First submitted 2022-04-16; First posted 2022-04-22 (Actual); Results first posted 2025-08-19 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Relative Energy Deficiency in Sport
Keywords: Bone metabolism; Endurance exercise; Low energy availability; Jump training
MeSH Terms: conditions — Relative Energy Deficiency in Sport

STUDY DESIGN:
Intervention Model Description: Randomized crossover study design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Endurance and Jumping Exercises (Experimental): 5 days of endurance treadmill running and 5 sets of 10 jumping exercises
  Interventions: Behavioral: Impact Load Exercises
- Endurance Exercise Only (Active Comparator): 5 days of endurance treadmill running
  Interventions: Behavioral: No Impact Load Exercises

INTERVENTIONS:
Behavioral: Impact Load Exercises — Participants will complete 50-65 min running protocol on treadmill and 5 sets of 10 jumping exercises for 5 consecutive days. Participants will also be provided all meals and snacks to induce a energy-restricted state for the 5-day period.
  Arms: Endurance and Jumping Exercises
Behavioral: No Impact Load Exercises — Participants will complete only a 50-65 min running protocol on treadmill for 5 consecutive days. Participants will also be provided all meals and snacks to induce a energy-restricted state for the 5-day period.
  Arms: Endurance Exercise Only

SUMMARY:
This study is a randomized, cross-over intervention study that will evaluate the effect of brief, high-impact loading exercises on biomarkers of bone metabolism in energy-restricted female runners. Volunteers will complete two 5-day experimental conditions in a randomized order separated by one menstrual cycle (approximately 3 weeks). Experimental conditions will include a dietary intervention of energy intake equal to 30 kcal/kg of fat-free mass/d using controlled diets and an exercise intervention of daily treadmill running with or without an additional 50 impact loading exercises.

DETAILED DESCRIPTION:
Many long-distance runners struggle to consume enough calories each day to match the number of calories they are burning during exercise and as part of daily living. Undereating for long periods of time is a serious concern because it can have negative effects on general health and sports performance. One of these long-term consequences is related to bone health. With undereating, bone can start to be broken down faster than it can be rebuilt. Even though it can take months, and even years, for bone to be seriously affected, this may lead to weak and brittle bones later in life, if it is left untreated. Typically, athletes are recommended to increase the number of calories they eat to prevent negative health concerns. However, not all athletes may be willing or able to increase their calories based on their performance goals, nutrition knowledge, or concerns with food security. This means that alternative strategies need to be investigated to counteract the negative effects of undereating on bone health. This study proposes to evaluate the effect of adding short bouts of high-impact jumping exercises to typical endurance training to promote healthy bone metabolism. This will specifically involve completing two phases of a supervised treadmill run and consuming a reduced-calorie diet (provided by the research team) on 5 consecutive days. In addition, one of the phases will include performing 5 sets of 10 jumping exercises on 5 consecutive days in addition to the treadmill run. Results of the study will serve as an important first step in helping exercise and medical professionals understand more about how to protect and manage the bone health of female long-distance runners.

ELIGIBILITY:
Inclusion Criteria:

* Females runners with regular menstrual cycles, not using contraceptives
* Body Mass Index between 18.5-30.0 kg/m2
* Weight stable (+/- 2 kg) for 6 months
* VO2max of ≥35 ml/kg/min
* Willing to consume provided meals and snacks

Exclusion Criteria:

* Low Energy Availability in Females Questionnaire (LEAF-Q) score ≥8
* Menstrual disturbances measured by progesterone and self-report
* Using contraceptives (oral contraceptives, injections, intrauterine device, etc.)
* Low Bone Mineral Density (z-score < -1)
* Routine engagement in mechanical loading exercises
* History of fracture in the previous 6 months
* Recent recovery (within the last 12 months) or still in recovery after eating disorder diagnosis
* Medication use that could affect bone metabolism (e.g., corticosteroids, anticonvulsants, heparin, gonadotropin-releasing hormone agonists)
* Pregnancy or lactation
* Abnormal thyroid-stimulating hormone levels

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2022-08-24 (Actual); Primary Completion 2024-01-23 (Actual); Study Completion 2024-04-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Enette Larson-Meyer, PhD, Principal Investigator — Virginia Polytechnic Institute and State University (Virginia Tech)
Locations (1):
- Virginia Polytechnic Institute and State University, Blacksburg, Virginia, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 38 individuals were screened for eligibility between August 2, 2022 and October 13, 2023 in Southwest Virginia.
Pre-assignment Details: 14 of 38 participants were randomized. Of those not randomized, 17 did not meet inclusion criteria and 7 declined to participate.
Groups:
- RUN, Then RUN+J: Participants first completed a 5-day period of energy restriction while running on the treadmill every day (RUN). After a washout period of at least one menstrual cycle, they then completed another 5-day period of energy restriction while running on the treadmill daily in addition to completing 5 sets of 10 jumping exercises each day (RUN+J).
- RUN+J, Then RUN: Participants first completed a 5-day period of energy restriction while running on the treadmill and completing 5 sets of 10 jumping exercises each day (RUN+J). After a washout period of at least one menstrual cycle, they then completed another 5-day period of energy restriction while only running on the treadmill each day (RUN).
Period: First Intervention (5 Days)
Arm/Group | RUN, Then RUN+J | RUN+J, Then RUN
Started | 7 | 7
Completed | 6 | 7
Not Completed | 1 | 0
Period: Washout (One Menstrual Cycle, ~21 Days)
Arm/Group | RUN, Then RUN+J | RUN+J, Then RUN
Started | 6 | 7
Completed | 6 | 5
Not Completed | 0 | 2
Period: Second Intervention (5 Days)
Arm/Group | RUN, Then RUN+J | RUN+J, Then RUN
Started | 6 | 5
Completed | 5 | 5
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | RUN, Then RUN+J | RUN+J, Then RUN | Total
Number analyzed (Participants) | 6 | 7 | 13
Age, Continuous [Mean (Standard Deviation); unit: Years] | 25.3 (4.2) | 26.9 (3.6) | 26.2 (3.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 7 | 13
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 5 | 5 | 10
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Bone Remodeling Biomarker - N-terminal Propeptide of Type 1 Procollagen
Description: Plasma N-terminal propeptide of type 1 procollagen (PINP) was collected from fasted blood samples drawn before and after each 5-day intervention. The enzyme-linked immunosorbent assays (ELISA) were performed on all samples upon study completion.
Time Frame: 10-minute blood draw in laboratory; samples assessed on intervention day 0 and day 6
Population: Only participants who completed the entire intervention period were included in the analysis.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Endurance and Jumping Exercises (RUN+J): Participants who completed 5 days of endurance treadmill running in addition to 50 high-impact jumping exercises daily.
- Endurance Exercise Only (RUN): Participants who completed 5 days of endurance treadmill running daily without any additional impact exercise.
Arm/Group | Endurance and Jumping Exercises (RUN+J) | Endurance Exercise Only (RUN)
Number analyzed (Participants) | 12 | 11
ng/mL | -3.1 (5.7) | 1.1 (7.2)
Statistical Analysis 1: Comparison: Endurance and Jumping Exercises (RUN+J) vs Endurance Exercise Only (RUN); Null hypothesis is that there was no difference in change of PINP between RUN and RUN+J; Test type: Superiority; p = 0.246, Mixed Models Analysis

2. Primary Outcome: Change in Bone Remodeling Biomarker - C-terminal Telopeptide of Type 1 Collagen (CTX)
Description: Serum C-terminal telopeptide of type 1 collagen (CTX) was collected from fasted blood samples drawn before and after each 5-day intervention. The enzyme-linked immunosorbent assays (ELISA) were performed on all samples upon study completion.
Time Frame: 10-minute blood draw in laboratory; samples assessed on intervention day 0 and day 6
Population: Only participants who completed the entire intervention period were included in the analysis.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Endurance and Jumping Exercises (RUN+J) | Endurance Exercise Only (RUN)
Number analyzed (Participants) | 12 | 11
ng/mL | 0.04 (0.09) | 0.04 (0.12)
Statistical Analysis 1: Comparison: Endurance and Jumping Exercises (RUN+J) vs Endurance Exercise Only (RUN); Null hypothesis is that there was no difference in change of CTX between RUN and RUN+J; Test type: Superiority; p = 0.714, Mixed Models Analysis

3. Primary Outcome: Change in Blood Metabolic Marker - Parathyroid Hormone
Description: Parathyroid hormone levels were measured from fasted blood samples collected before and after each 5-day intervention. The enzyme-linked immunosorbent assays (ELISA) were performed on all samples upon study completion.
Time Frame: 10-minute blood draw in laboratory; samples assessed on intervention day 0 and day 6
Population: Only participants who completed the entire intervention period were included in the analysis.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Endurance and Jumping Exercises (RUN+J) | Endurance Exercise Only (RUN)
Number analyzed (Participants) | 12 | 11
pg/mL | 3.3 (6.1) | -1.0 (11.8)
Statistical Analysis 1: Comparison: Endurance and Jumping Exercises (RUN+J) vs Endurance Exercise Only (RUN); Test type: Superiority; p = 0.309, Mixed Models Analysis

4. Primary Outcome: Change in Blood Metabolic Marker - Insulin-like Growth Factor-1
Description: Insulin-like growth factor-1 (IGF1) concentration was measured from fasted blood samples collected before and after each 5-day intervention. The enzyme-linked immunosorbent assays (ELISA) were performed on all samples upon study completion.
Time Frame: 10-minute blood draw in laboratory; samples assessed on intervention day 0 and day 6
Population: Only participants who completed the entire intervention period were included in the analysis.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Endurance and Jumping Exercises (RUN+J) | Endurance Exercise Only (RUN)
Number analyzed (Participants) | 12 | 11
ng/mL | -11.4 (10.3) | -8.0 (6.3)
Statistical Analysis 1: Comparison: Endurance and Jumping Exercises (RUN+J) vs Endurance Exercise Only (RUN); Null hypothesis is that there was no difference in change of IGF1 between RUN and RUN+J; Test type: Superiority; p = 0.308, Mixed Models Analysis

5. Secondary Outcome: Change in Ferritin
Description: Fasted serum ferritin was measured before and after each 5-day intervention period.
Time Frame: 10-minute blood draw in laboratory; samples assessed on intervention day 0 and day 6
Population: Only participants who completed the entire intervention period were included in the analysis.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Endurance and Jumping Exercises (RUN+J) | Endurance Exercise Only (RUN)
Number analyzed (Participants) | 12 | 11
ng/mL | 4.1 (11.3) | 11.4 (11.5)
Statistical Analysis 1: Comparison: Endurance and Jumping Exercises (RUN+J) vs Endurance Exercise Only (RUN); Null hypothesis is that there was no difference in change of ferritin between RUN and RUN+J; Test type: Superiority; p = 0.207, Mixed Models Analysis

ADVERSE EVENTS:
Time Frame: One week for each intervention.
Description: Safety Population included all participants who were consuming energy-restricted diets during the intervention period.
Groups:
- Endurance and Jumping Exercise (RUN+J): Participants completed 5 consecutive days of exercise consisting of daily endurance treadmill running and 50 high-impact jumping exercises. The 5-day period was under a controlled energy availability condition of 15 kcal/kgFFM/day.
- Endurance Exercise Only (RUN): Participants completed 5 consecutive days of daily endurance treadmill running without any additional impact exercise. The 5-day period was under a controlled energy availability condition of 15 kcal/kgFFM/day.
Arm/Group | Endurance and Jumping Exercise (RUN+J) | Endurance Exercise Only (RUN)
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/10
Other Adverse Events (participants affected / at risk) | 0/12 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-09-11): https://cdn.clinicaltrials.gov/large-docs/00/NCT05341700/Prot_SAP_000.pdf